CLINICAL TRIAL: NCT03101475
Title: Phase II of Immunotherapy Plus Local Tumor Ablation (RFA or Stereotactic Radiotherapy) in Patients With Colorectal Cancer Liver Metastases
Brief Title: Synergism of Immunomodulation and Tumor Ablation
Acronym: ILOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1560-GITCG; 2017-001375-22 (EudraCT Number)
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Colorectal Cancer; Liver Metastases; Durvalumab; Tremelimumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — durvalumab; tremelimumab; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immunotherapy + local tumor ablation (Experimental): Patients with unresectable colorectal liver metastases which show at least stable disease or partial remission after 4-6 months will receive treatment with durvalumab and tremelimumab plus local tumor ablation (Radiofrequency ablation RFA or Sterotactic body radiation therapy SBRT) of selected liver lesions, followed by maintenance treatment with durvalumab.
  Interventions: Drug: Durvalumab (MEDI4736); Drug: Tremelimumab; Radiation: Sterotactic body radiation therapy (SBRT); Other: Radiofrequency ablation (RFA)

INTERVENTIONS:
Drug: Durvalumab (MEDI4736) — Durvalumab (MEDI4736) 1500mg Q4W in combination with tremelimumab for up to 4 doses/cycles, followed by durvalumab (MEDI4736) 1500mg Q4W for up to a maximum of 8 months with the last administration on week 48 unless there is unacceptable toxicity.
Drug: Tremelimumab — Tremelimumab (75 mg IV Q4W) in combination with durvalumab (MEDI4736) (1500mg Q4W) for up to 4 doses/cycles
Radiation: Sterotactic body radiation therapy (SBRT) — delivered in 3 fractions of 10 Gy over 1 week starting 8 to 14 days after first dose of immunotherapy
Other: Radiofrequency ablation (RFA) — performed percutaneously under CT, MRI or sonographic guidance 8 to 14 days after start of immunotherapy

SUMMARY:
This is a single-arm, open-label, multi-center early phase II study. This proof of concept study will investigate whether the combined use of local tumor ablation/radiation plus immunomodulating drugs may induce a significant immune response in patient with incurable liver metastases from colorectal cancer (CRC) (+/- limited extrahepatic disease) being stable or in partial remission after completion of 4-6 months first line systemic therapy.

The primary objective of the study is to show an overall response rate of lesions not treated by ablation/radiotherapy including the extrahepatic lesions (according to iRECIST criteria) higher than 10%. With the continuation of first line systemic treatment, no further responses are expected.

Secondary objectives are:

* To establish the feasibility and safety of the combined treatment modalities;
* To study the impact of the local technique (RFA/Radiotherapy) on the results;
* To investigate biomarkers to predict response to the combined treatment

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically confirmed CRC
* Patients with CRC liver metastases, with or without extrahepatic disease, in which curative treatment is not possible by resection and or local ablation/radiotherapy.
* ≥ 18 years of age at time of study entry
* WHO performance status 0 to 1
* Body weight > 30kg
* Measurable disease according to RECIST 1.1
* Stable disease or partial remission by RECIST 1.1 criteria after at least 3 months systemic therapy for CRC. Patients following first- or second-line treatment are eligible. Note: if patient receives maintenance treatment after the first line treatment, she/he remains eligible for this study
* Complete responders or partial responders with a 80% or more decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions following systemic therapy, taking as reference the sum of diameters from baseline scan prior to initiation of first line therapy are excluded as well as patients with almost complete cystic degeneration of liver metastases. Note: The interval between last dose of systemic treatment and first dose of study drugs must be maximum 8 weeks (in case bevacizumab was administered as part of the systemic treatment, a minimum 21 days wash out period is required from last administration to planned local ablative treatment initiation).
* Liver metastases amenable to ablation or stereotactic radiotherapy (SBRT) at completion of systemic therapy:
* For SBRT: allowing a total ablated volume of at least 25 cm3 and a maximum of 40 cm3 with a maximum of two lesions treated with SBRT
* For RFA: allowing a total ablated volume of at least 25 cm3 and a maximum advised volume of 120 cm3
* At least two measurable liver metastases, or at least 1 measurable liver metastasis and 1 measurable extrahepatic lesion should remain untreated by ablation or SBRT to allow response monitoring according to RECIST 1.1 and iRECIST.
* Limited extra hepatic disease is allowed, including up to 2 extra hepatic metastatic sites, either lung, abdominal, pelvis, bone, or localized lymph node metastases. Each will be counted separately as one site. So, two abdominal lesions will be counted as 1 extra-hepatic site; one lung and one abdominal lesion will be counted as two sites. Individual extrahepatic lesions should be ≤ 5 cm.
* Availability of tumor sample for biomarkers testing (MSI, PDL-1, etc) (archival tissue from primary tumor or biopsy)
* Adequate normal organ and marrow function before initial systemic treatment as well as at baseline as defined below:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
* Platelet count ≥ 100 x 109/L (>100,000 per mm3)
* Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* AST (SGOT)/ALT (SGPT) ≤ 5 x institutional upper limit of normal
* Creatinine ≤ 1.5 x institutional ULN or measured or calculated creatinine clearance >40 mL/min by the Cockcroft-Gault formula (Appendix E)
* Hemoglobin ≥ 9.0 g/dL at baseline
* Patient with following medical conditions are eligible:
* Patients with vitiligo or alopecia
* Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients with celiac disease controlled by diet alone
* No history of another malignancy or a concurrent malignancy. Exceptions include patients who have been disease-free for 5 years, or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ.
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the first dose of study treatment. Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrhoeic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy the last study treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:
* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomized partner
* Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient) Note: please refer to Appendix J for Clinical Trial Facilitation Group (CTFG) guidelines.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment, from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations

EXCLUSION CRITERIA

* Patients with known brain metastases or history of leptomeningeal carcinomatosis
* Hilar liver lesions close to central bile ducts to be treated by RFA
* Prior treatment:
* History of radiation therapy of the liver, upper abdomen or lower thorax
* History of radioembolization of the liver
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of durvalumab and tremelimumab.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab, a CTLA-4 including tremelimumab or other checkpoint inhibitors or other immune therapy during the last 12 months
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab and tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid, or steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
* Any unresolved toxicity NCI CTCAE v 4.0 Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory pulmonary disorders, interstitial lung disease, inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab, tremelimumab or any excipient
* Uncontrolled intercurrent illness including, but not limited to:
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Active peptic ulcer disease or gastritis
* Liver cirrhosis CHILD B+, C (Appendix I)
* Active bleeding diatheses
* History of primary immunodeficiency
* Cardiac disorders:
* Symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
* Female patients who are pregnant or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial Blood donation: Subjects should not donate blood while participating in this study, or for at least 90 days following the last infusion of durvalumab or tremelimumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Best overall immune response rate (iBOR) of lesions not treated by ablation/radiotherapy including the extrahepatic lesions according to iRECIST (with response confirmation) | 36 months from first patient in
  The statistical design is based on the assumption that the continuation of first line systemic treatment would result in nearly no further response translating into a response rate of 0 to 5% at maximum in the enrolled patient's population. A response rate of 10% in the experimental arm (local treatment + immunotherapy) will be judged too low to justify this combined approach. On the contrary, a response rate of 25% will be judged very promising. An optimal Simon's two-stage design will be used for the rejection of a 10% or less iBOR rate

SECONDARY OUTCOMES:
Best overall immune response rate of liver lesions not treated with local therapy according to iRECIST (with response confirmation) | 36 months from first patient in
  iBOR rate of liver lesions not treated with local therapy according to iRECIST (with response confirmation) will be displayed (point estimate) with their exact two-sided 95% confidence intervals.
Best overall response rate of lesions not treated by ablation/radiotherapy including or not the extrahepatic lesions according to RECIST v1.1 (with response confirmation) | 36 months from first patient in
  BOR rate of lesions not treated by ablation/radiotherapy including or not the extrahepatic lesions according to RECIST v1.1 (with response confirmation) will be displayed (point estimate) with their exact two-sided 95% confidence intervals.
Response duration | 54 months from first patient in
  Response duration will be presented using the median, range (minimum, maximum) and inter-quartile range as well as the mean and standard deviation.
Stable disease duration | 54 months from first patient in
  Stable disease duration will be presented using the median, range (minimum, maximum) and inter-quartile range as well as the mean and standard deviation.
Progression free survival according to iRECIST and to RECIST v1.1 | 54 months from first patient in
  Progression free survival according to iRECIST and RECIST v1.1 curve will be estimated using the Kaplan-Meier technique. Medians will be displayed with their two-sided 95% confidence intervals.
Overall survival | 54 months from first patient in
  Overall survival curve will be estimated using the Kaplan-Meier technique. Medians will be displayed with their two-sided 95% confidence intervals.
Safety: Safety analyses will be performed on the Safety population. The worst toxicity grade per patient over the treatment period according to the CTCAE criteria version 4.0 will be displayed. | 54 months from first patient in
  Safety analyses will be performed on the Safety population. The worst toxicity grade per patient over the treatment period according to the CTCAE criteria version 4.0 will be displayed.

CONTACTS AND LOCATIONS:
Overall Officials: Theo Ruers, Study Chair — The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, The Netherlands; Jenny Seligmann, Study Chair — Leeds Teaching Hospitals NHS Trust - St. James's University Hospital
Locations (10):
- Medical University Vienna - General Hospital AKH, Vienna, Austria
- Institut Bergonie, Bordeaux, France
- Germany (2):
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum Leipzig-Ambulanzen/Sprechstunden, Leipzig
- Netherlands (2):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Radboud University Medical Center Nijmegen, Nijmegen
- Karolinska University Hospital - Karolinska Institutet - Danderyds Hospital, Stockholm, Sweden
- Switzerland (3):
  - Inselspital, Bern
  - Hôpitaux universitaires de Genève - HUG - site de Cluse-Roseraie, Geneva
  - UniversitaetsSpital Zurich, Zurich